CLINICAL TRIAL: NCT06431828
Title: Efficiency of a Clinical Process Based on Remote Review of Symptoms in Patients With an Implantable Diagnostic Holter.
Brief Title: Remote Symptom Review in Patients With Implantable Diagnostic Holter
Acronym: BIOMONI-DIG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Andres Iñiguez Romo (Other)
Collaborators: Fundacin Biomedica Galicia Sur (Other); Fundacion Investigacion Interhospitalaria Cardiovascular (Other)
Responsible Party: Sponsor-Investigator, Andres Iñiguez Romo, Head of Cardiology, Fundacin Biomedica Galicia Sur
Organization: Fundacin Biomedica Galicia Sur (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: FF088
Record Dates: First submitted 2024-05-08; First posted 2024-05-29 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Atrial Fibrillation; Syncope; Bradycardia; Arrythmia
Keywords: Implantable loop recorder; Arrythmia; Atrial Fibrillation; Home Monitoring
MeSH Terms: conditions — Atrial Fibrillation; Syncope; Bradycardia; Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Homemonitoring + APP (Experimental): The patients receive the usual standard treatment with remote holter monitoring along with an app for the notification of adverse events.
  Interventions: Other: APP
- Homemonitoring (No Intervention): The patients receive the usual standard treatment with remote holter monitoring

INTERVENTIONS:
Other: APP — The patients will download an app through which they will be able to report adverse events related to their cardiovascular health.
  Arms: Homemonitoring + APP

SUMMARY:
To study the clinical and organizational benefit of implementing a methodology for monitoring patients receiving an implantable diagnostic BIOMONITOR III holter and successive models, consisting of remote review of alerts sent by the device via the HOME MONITORING remote monitoring platform and the transmission of relevant patient symptoms through the use of a specific application installable on the patient's phone. The efficiency of this methodology will be compared with a control group consisting of monitoring through the usual clinical practice of the hospital.

DETAILED DESCRIPTION:
Population of patients: Patients over 18 years old who require the implantation of an implantable diagnostic holter due to indications of syncope or atrial fibrillation, and who are willing to use an application installed on their phone to telematically send clinical symptoms that may occur during the active study period.

Design: Clinical, randomized, prospective, single-center study.

Investigational Device: BIOMONITOR III implantable cardiac holter and successive models with HOMEMONITORING remote monitoring system for constant monitoring of patient's cardiac signals. Installation of the Patient APP on the patient's phone for symptom transmission.

Overall Objective: To study the clinical and organizational benefit of implementing a methodology for monitoring patients receiving an implantable diagnostic BIOMONITOR III holter and successive models, consisting of remote review of alerts sent by the device via the HOME MONITORING remote monitoring platform and the transmission of relevant patient symptoms through the use of a specific application installable on the patient's phone. The efficiency of this methodology will be compared with a control group consisting of monitoring through the usual clinical practice of the hospital.

ELIGIBILITY:
Inclusion Criteria:

* Patients indicated for implantation of a subcutaneous implantable holter due to syncope or cryptogenic stroke (atrial fibrillation detection)
* Patients over 18 years old.
* Patients who consent to the installation of a patient application for telematic submission of patient-related symptoms.
* Patients capable of using the patient application.

Exclusion Criteria:

* Patients over 80 years of age or, failing that, not able to use an application to send their symptoms.
* Life expectancy of less than 12 months for any reason.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-04-22 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
TIME FRAME | one year
  Time from the first alert by Home Monitoring of the implantable holter to the clinical diagnosis according to the patient's clinical indication.

SECONDARY OUTCOMES:
Number of in-person visits in each group | one year
  Number of in-person visits in each group
Incidence remote transmissions activated by patient indication | one year
  Number of remote transmissions activated by patient indication
Rate of false positives | one year
  Number of false positives, according to physician's diagnosis.
Rate of symptoms sent by the patient | one year
  Number of false positives (according to physician's diagnosis)
Rate of symptoms sent by the patient that correspond to remote alerts sent by the patient | one year
  Rate of symptoms sent by the patient that correspond to remote alerts sent by the patient (e.g., the symptom corresponds to a detected arrhythmia)
Rate of symptoms not corresponding to detected arrhythmias | one year
  Rate of symptoms not corresponding to detected arrhythmias(e.g., the symptom corresponds to a detected arrhythmia)
Number of new non-cardiac clinical diagnoses discovered thanks to the symptoms sent by the patient. | one year
  Number of new non-cardiac clinical diagnoses discovered thanks to the symptoms sent by the patient.corresponds to a detected arrhythmia
Efficacy of implementing a clinical process based on remote monitoring of patient symptoms | one year
  Change in patient interaction with the physician - fewer calls/visits to the hospital.
Qualitative Patient Objectives | one year
  Measured through a satisfaction survey on the use or non-use of the patient application to telematically send their symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Andrés Iñiguez Romo, MD, phD, Study Chair — Servicio Galego de Saude
Locations (1):
- Hospital Álvaro Cunqueiro, Vigo, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gupta N, Yang J, Reynolds K, Lenane J, Garcia E, Sung SH, Harrison TN, Solomon MD, Go AS; KP-RHYTHM Study Group. Diagnostic Yield, Outcomes, and Resource Utilization With Different Ambulatory Electrocardiographic Monitoring Strategies. Am J Cardiol. 2022 Mar 1;166:38-44. doi: 10.1016/j.amjcard.2021.11.027. Epub 2021 Dec 23. PMID 34953575
- [Result] Sharma AN, Baranchuk A. Ambulatory External Electrocardiography Monitoring: Holter, Extended Holter, Mobile Cardiac Telemetry Monitoring. Card Electrophysiol Clin. 2021 Sep;13(3):427-438. doi: 10.1016/j.ccep.2021.04.003. Epub 2021 Jul 8. PMID 34330370
- [Result] Varma N, Epstein AE, Schweikert R, Michalski J, Love CJ; TRUST Investigators. Role of Automatic Wireless Remote Monitoring Immediately Following ICD Implant: The Lumos-T Reduces Routine Office Device Follow-Up Study (TRUST) Trial. J Cardiovasc Electrophysiol. 2016 Mar;27(3):321-6. doi: 10.1111/jce.12895. Epub 2016 Jan 27. PMID 26661687